CLINICAL TRIAL: NCT00544518
Title: Impact of Benfluorex Versus Metformin on Glucose Control and Insulin Secretion in Chinese Type 2 Diabetic Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: Shandong Xinhua Pharmaceutical Company Limited in China (Unknown); Beijing Haijinge medicine Science-tech CO.,LTD(CRO) (Unknown); Center for Drug Clincal Reserch Shanghai University of TCM (Other); Beijing Army General Hospital (Other Government); Bethune International Peace Hospital (Other); The People's Hospital of Hebei Province (Other); Second Hospital of Jilin University (Other)
Responsible Party: the clinical trial center, Xijing Hospital, The fourth military medical university
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: bfls071012
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; Benfluorex; Metformin; insulin secretion; glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; benfluorex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental)
  Interventions: Drug: benfluorex
- 1 (Active Comparator)
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: metformin — 2 tablets with breakfast and dinner for the first four weeks, if necessary, increase 2 tablets with noon for the next time
  Arms: 1
Drug: benfluorex — 2 tablets with breakfast and dinner for the first four weeks, if necessary, increase 2 tablets with noon for the next time, one of 2 tablets is dummy tablet.
  Arms: 2

SUMMARY:
Objective--- Benfluorex may have effects on the glucose control in type 2 diabetes while it improves hyperlipidemia. We sought to compare the impacts of benfluorex versus metformin on glucose control and insulin secretion in Chinese type 2 diabetic patients.

Research design and methods---a 16-week, double-blind, multiple centers, random parallel controlled study is designed to compare the impact of benfluorex (150-450mg/day, provided by Shandong Xinhua Pharmaceutical Company Limited in China) on glucose control, insulin secretion and its safety with metformin in type 2 diabetic patients. 240 type 2 diabetic patients are to be recruited to receive benfluorex or metformin(1:1). HbA1c, plasma lipid level, insulin and glucose at 0', 30', 120' after a standard meal will be measured before and after treatment, while fasting and postprandial glucose measured 4 times regularly. The change of HbA1c from baseline to the end of treatment will taken as main efficacy criterion, as the changes of fasting and after standard meal glucose and insulin level and plasma lipid level will be taken as secondary criteria. All patient will be given safety monitor at prior and post treatment. Data management and statistical analysis will adopt DAS for Clinical Trial 2.0.

DETAILED DESCRIPTION:
During the whole study, patients meet a physician on a regular basis. Safety is assessed by adverse event spontaneous reporting、physical examination、recording of vital signs、laboratory tests and electrocardiogram at baseline and 16 week . Blood samples are collected for centralized measure of HbA1C and fasting serum insulin(FSI)、PSI1/2、PSI2 after an overnight fast in all patients,Body weight, supine and standing blood pressures and heart rate are measured at each clinical visit. Adverse events are rated as mild, moderate or severe by the investigators and assessed for any causal relationship to the study drugs. Patients are entitled to interrupt the treatment at any time during the study, and investigators can withdraw patients, in particular if they are inadequately controlled.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the study, participants will be；① Antidiabetic drugs naïve Type 2 diabetes mellitus（WHO standard） with diet control more than 2 weeks; ②or diagnosed Type 2 diabetes mellitus with no oral antidiabetic drugs more than 6months; ③or Type 2 diabetes mellitus treated with insulin secretagogues more than 1 month; all patients have HbA1c between 7.0-10.0% and fasting glucose between 7.0mmol/L～13.0mmol/L.
* Ages Eligible for Study: 18 Years --70 Years, Genders:Both
* BMI: 23～40kg/m2
* No using insulin before 3 months
* Consent to do birth control to Women of child-bearing age
* Volunteer to join and sign Information consent form

Exclusion Criteria:

* Patients with ketoacidosis、hyperglycemic hyperosmolar syndrome.
* Patients with severe diabetic complications
* Patient with acute cardiovascular diseases，acute cerebrovascular diseases，with Vitamin B12、folic acid and iron deficiency，with severe trauma or surgery，severe infection diseases.
* Allergy to benfluorex or metformin
* ALT、AST> 2 times of upper normal limit，Cr> upper normal limit.
* Having used benfluorex within 3 months before recruiting.
* Patients accepting steroid hormones or malignant tumor treatment
* Patients with drug abuse or bibulous history.
* Patients with severe unconscious low blood glucose history，severe mental illness history and family history
* Severe hypertensive patients（SBP>160 mmHg，DBP>95mmHg）
* Patient with pancreas diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-09 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
The change of HbA1c from baseline to the end of treatment | 16 weeks

SECONDARY OUTCOMES:
the changes of fasting and after standard meal glucose and insulin level and plasma lipid level | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ji qiuhe, Ph.D, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- XiJing hospital of Fourth Military Medical University, Xi’an, Shanxi, China